CLINICAL TRIAL: NCT05953155
Title: Effectiveness of YOga in Patients with Chronic Low BACK Pain and Poor PROgnosis (YOBACK-PRO Trial): a Randomized Controlled Trial
Brief Title: YOga for Patients with Chronic BACK Pain and Poor PROgnosis
Acronym: YOBACK-PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Rafael Zambelli Pinto, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 57028022.0.0000.5149
Record Dates: First submitted 2023-07-12; First posted 2023-07-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain; Chronic Low-back Pain; Back Pain; Back Pain Lower Back Chronic
Keywords: low back pain; chronic low back pain; yoga; poor prognosis
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): The control group will be invited to attend 3 educational classes. In these sessions, participants will receive evidence-based information about self-management strategies and pain education.
  Interventions: Other: Control
- Yoga (Experimental): In addition to the invitation to attend the same 3 educational classes on evidence-based information about self-management strategies and pain education, the experimental group will participate in a 12-week, twice-weekly group-based yoga program.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Control — Each educational class will last for 1 hour and consists of evidence-based information about low back pain, including, for example, self-management strategies, pain education, reassurance and common misconceptions about back pain.
  Arms: Control
Other: Yoga — Participants in the intervention group will receive, in addition to the educational classes, a course of yoga program led by certified yoga instructors. The program consists of a 60-min group session with up to 10 participants, delivered twice a week for 12 weeks.
  Arms: Yoga

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of yoga for patients with chronic low back pain and high risk of poor prognosis. The main question it aims to answer is:

- In patients with back pain and high risk of poor prognosis, what is the effectiveness of yoga plus education on reducing pain and disability compared to a control group receiving education alone?

A total of 110 patients with chronic low back pain and classified as high risk of poor prognosis according to the Orebro Musculoskeletal Pain Screening Questionnaire (i.e. score ≥ 50 points out of 100) will be recruited for this study. Participants will be randomized into two groups: yoga and control. The yoga group will receive a 3-month course of yoga program consisting of two sessions per week and 3 educational classes. The control group will receive 3 educational classes over a 12-week period. Outcome measures will be assessed at baseline, at post-intervention (i.e. 3-months post randomization) and at 6-month follow up (i.e. 6-months post randomization).

ELIGIBILITY:
Inclusion Criteria:

* report chronic nonspecific LBP, defined as pain and discomfort localized below the costal margin and above the inferior gluteal folds, with or without leg pain and of at least 3 months' duration.
* score ≥ 50 points (out of 100) in the Orebro Musculoskeletal Pain Questionnaire.
* have an average back pain intensity of 3 points or more on a 0-10 numerical pain rating scale.

Exclusion Criteria:

* serious spine pathology (e.g. tumors, fractures, and inflammatory diseases).
* nerve root compromise (i.e. at least 2 of the following signs: weakness, reflex change, or sensation loss associated with the same spinal nerve).
* previos spinal surgery.
* pregnancy or having given birth within the previous 3 months.
* any medical condition that prevented being physically active (e.g., serious cardiovascular, kidney or neurological diseases).
* any other musculoskeletal condition that may affect activity and movement participation in a Yoga program during the last year.
* not currently receiving other physical activity-based intervention (e.g., Pilates, physical therapy, aquatic exercise).
* inadequate Portuguese literacy for the study's questionnaires and instructions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Disability | Post-intervention (i.e. 3 months after randomisation)
  Roland Morris Disability Questionnaire (RMDQ) (0-24 scale)

SECONDARY OUTCOMES:
Disability | 6 months after randomisation
  Roland Morris Disability Questionnaire (RMDQ) (0-24 scale)
Pain intensity | Post-intervention (i.e. 3 months after randomisation) and at 6-month follow-up
  Numerical Rating Scale for Pain assessment (NRS) (0-10 scale)
Quality of life | Post-intervention (i.e. 3 months after randomisation) and at 6-month follow-up
  EuroQol Visual Analogue Scale (EQ-VAS) (0-100 scale)
Depressive symptoms | Post-intervention (i.e. 3 months after randomisation) and at 6-month follow-up
  Center for Epidemiological Studies - Depression (CES-D) (0-60 scale)
Pain self-efficacy | Post-intervention (i.e. 3 months after randomisation) and at 6-month follow-up
  Pain Self-Efficacy Questionnaire (PSEQ) (0-60)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Z Pinto, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- IPSEMG - Instituto de Previdência dos Servidores do Estado de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
The data of this study will be available from the principal investigator upon reasonable request.

REFERENCES:
- [Derived] Nunes SM, Rizzo RR, Franco MR, Ferreira FR, Barros LJG, Maciel IT, Santos RL, Nascimento RR, Couto AJ, Quaresma LS, Fontes RM, Ferreira EMR, Maher CG, McAuley JH, Pinto RZ. Efficacy of YOga in people with chronic non-specific low BACK pain and poor PROgnosis (YOBACK-PRO): protocol for a randomised clinical trial. BMJ Open. 2026 Jan 28;16(1):e112982. doi: 10.1136/bmjopen-2025-112982. PMID 41605601